CLINICAL TRIAL: NCT03839732
Title: Calcify2D: Assessment of Observer Variability of a New Software for the Quantitative Evaluation of Abdominal Aortic Calcifications, Vertebral Morphometry and Their Relationships in Fragile Patients, Compared to Current Visual Scoring Methods
Brief Title: Observer Variability in Scoring Abdominal Aortic Calcifications and Vertebral Morphometry
Acronym: CALCIFY2D
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: CE AVEC 695/2018/Oss/IOR
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Vascular Calcification; Vertebral Fracture
Keywords: observer variability; kauppila score; quantitative vertebral morphometry; computer assisted procedure; abdominal aorta; lumbar spine
MeSH Terms: conditions — Vascular Calcification; Spinal Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vascular Calcification Group: Patients with prevalent vascular calcifications will be analysed to verify the intra- and inter-observer reliability of the score of abdominal aorta calcifications
  Interventions: Diagnostic Test: Score of abdominal aorta calcifications

INTERVENTIONS:
Diagnostic Test: Score of abdominal aorta calcifications — Radiographs showing VC will be used to assess whether the computer assisted VC scoring (primary objective) and Quantitative Vertebral Morphometry (QVM, limited to lumbar spine, secondary objective n.1) through the Calcify2D software are less variable with respect to the traditional visual scoring of VC and QVM.
  Other Names: Score of lumbar spine vertebral fractures

SUMMARY:
BACKGROUND In the context of a progressively aging population, monitoring the status of Vascular Calcifications (VC) and Vertebral Fractures (VF) over time would be of primary importance, as VC and VF are recognized to be hallmarks of severe cardiovascular events (hospitalization and/or death) and hip fractures respectively, and VF represent an under-diagnosed cause of progressive disability and pain on its own. Moreover, there is an acknowledged relationships between VC and VF.

However, data about the emergence/progression of VC and the emergence/worsening of VF over time are lacking. This is likely due to the absence of monitoring instruments for VC and VF that are both precise and easily accessible/applicable.

OBJECTIVE This study aims to define the observer variability of a new software developed by the study sponsor and collaborators, called Calcify2D. Calcify2D offers physicians a computer-assisted procedure to simultaneously score vascular calcifications at the abdominal aorta and lumbar vertebral fractures (according to Quantitative Vertebral Morphometry principles) based on a latero-lateral thoracolumbar spine radiography. Secondary aims are the validation of the scores obtained from latero-lateral thoracolumbar spine radiography with more invasive and/or costly gold-standard imaging modalities (Computed Tomography for VC, Magnetic Resonance for VF) that may have been acquired near-simultaneously to radiographs on the patients enrolled for the study.

STUDY DESIGN Not-for-profit monocentric observational study to be conducted on the diagnostic images of the thoracolumbar spine already collected at Istituto Ortopedico Rizzoli (IOR) within a previous interventional study.

Scoring of VC and VF will be performed by four clinicians from four relevant specialties, chosen among those who may often see VC and VF and are already familiar with the traditional scoring systems for both VC and VF (one radiologist and one spine orthopaedics from IOR, one nephrologist from the National Research Council and one internist from University of Padua).

Each clinician will assess all radiographs to score VC and QVM, both via computer assisted procedures and via traditional visual inspection. To avoid bias, an interval of at least one week will be left between the computer assisted and visual scoring. To define intra-observer variability (i.e. repeatability), the whole dataset will be re-assessed three times.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in a previous interventional study (VTP vs KYPHO) of the sponsor.
* Availability of diagnostic images (Dorso-lumbar radiographies taken in L-L projection).
* Rx images will be screened for the presence of VC, retaining only those showing VC.
* Informed consent obtained prior to any study analysis-evaluation.

Exclusion Criteria:

* Images showing severe artefacts (usually due to presence of metallic devices) that alter the grayscale range and hinder correct identification of VC and vertebral fractures

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients that were included in a previous interventional trial of the sponsor institution aimed to compare the effectiveness of vertebroplastic and kyphoplastic augmentations of the throracolumbar spine. The choice of this population was driven by previous reports on similar populations stating a high prevalence of vascular calcifications.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Observer variability in scoring Vascular Calcification at the abdominal aorta | through study completion, 1 year at maximum
  Observer variability (repeatability and reproducibility) in the assessment of vascular calcifications at the abdominal aorta according to a widely adopted scoring system (Kauppila et al., 1997): comparison between computer assisted and visual scoring.

SECONDARY OUTCOMES:
Observer variability in scoring Vertebral Fractures at the lumbar spine | through study completion, 1 year at maximum
  Observer variability (repeatability and reproducibility) in the assessment of vertebral fractures in the lumbar spine according to Quantitative Vertebral Morphometry (Genant et al., 2000): comparison between computer assisted and visual scoring.
Accuracy of computer assisted VC score | through study completion, 1 year at maximum
  Accuracy of VC score computed by Calcify2D software will be tested against a gold standard CT-based score
Accuracy of computer assisted QVM | through study completion, 1 year at maximum
  Accuracy of QVM score computed by Calcify2D software will be tested for the detection of mild vertebral fractures against gold standard Magnetic Resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Schileo, Ph.D., Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT03839732/Prot_SAP_000.pdf